CLINICAL TRIAL: NCT07230015
Title: The Effectiveness of Combination of Motor Imagery and Vestibular Rehabilitation on Balance, Cognition, and Quality of Life in Patients With Multiple Sclerosis
Brief Title: Combined Motor Imagery and Vestibular Rehab for MS
Acronym: MIVR-MS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Gehad Salem Mohamed Mohamed Menshawi, PT, MSc (Cand.), Medipol University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E-10840098-202.3.02-1593
Record Dates: First submitted 2025-09-23; First posted 2025-11-17 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Multiple Sclerosis (MS) - Relapsing-remitting
Keywords: physical therapy; neurological rehabilitation; MS; Vestibular rehabilitation; Motor imagery; balance; QOL; Cognation; randomized control trial; physical therapy modalities; Physical therapy and rehabilitation; physical performance; Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis

STUDY DESIGN:
Intervention Model Description: This is a parallel group randomized controlled trial with two arms: an intervention group receiving motor imagery plus vestibular rehabilitation and a control group receiving conventional therapy only.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will not be informed of their group allocation. Due to the nature of the intervention, the investigator and care provider will be aware of the assignments, and the outcome assessments will also be conducted by the investigator."
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Motor Imagery + Vestibular Rehabilitation Group (Experimental): Participants receive a combined intervention of motor imagery and vestibular rehabilitation. Sessions last 55 minutes, including 5 min breathing warm-up, 20 min motor imagery training, 20 min vestibular exercises for balance and dizziness reduction, and 10 min cool-down/relaxation. The program aims to improve balance, cognitive function, and quality of life in patients with Multiple Sclerosis. Symptoms are monitored to avoid overexertion or symptom exacerbation.
  Interventions: Behavioral: Motor Imagery + Vestibular Rehabilitation group
- Conventional Group (Other): Participants receive conventional care for Multiple Sclerosis, including routine medical follow-up and standard physiotherapy if applicable. No specific motor imagery or vestibular rehabilitation exercises are administered. This group serves as a comparison to evaluate the effects of the experimental intervention.
  Interventions: Behavioral: Conventional therapy group

INTERVENTIONS:
Behavioral: Motor Imagery + Vestibular Rehabilitation group — This 8-week program, 3 sessions/week, 55- 60 min each, includes 4 steps:
  Warm-up (5 min): Breathing exercises progressing from basic diaphragmatic and pursed-lip breathing (weeks 1-2), light movement with breathing (weeks 3-4), to Inspiratory Muscle Training device (weeks 5-8).
  Motor Imagery (15 min): Foundational phase (weeks 1-2) imagining basic movements, skills building (weeks 3-4) with functional daily tasks, advanced phase (weeks 5-8) imagining complex tasks, environmental and cognitive challenges (e.g., sports, obstacle navigation, walking on uneven surfaces).
  Vestibular Rehabilitation (15 min): Foundational (weeks 1-2) gaze stabilization and static balance (VOR, VSR, VCR), dynamic balance and dual-task exercises (weeks 3-6), advanced functional balance and vestibular-cognition integration (weeks 7-8).
  Cool-down (10 min): Relaxation and symptom monitoring to prevent overexertion, dizziness, or fatigue.
  Arms: Motor Imagery + Vestibular Rehabilitation Group
Behavioral: Conventional therapy group — This 8-week program, 3 sessions/week, 55- 60 min each, includes:
  Warm-up: Seated/standing marching, neck and shoulder stretching.
  Strength & Functional Movements: Sit-to-stand, side leg raises, step-ups.
  Core & Upper Body: Bridge exercise, seated core activation, seated leg lifts, wall push-ups, seated shoulder press.
  Flexibility & Balance: Calf and hamstring stretches, spinal flexibility, single-leg stance, lunges, tandem walking.
  Cool-down: Deep breathing and gentle stretching.
  Arms: Conventional Group

SUMMARY:
This trial investigates the first combined use of motor imagery and vestibular rehabilitation in multiple sclerosis, aiming to evaluate their joint effect on balance, cognition, and quality of life.

DETAILED DESCRIPTION:
Multiple sclerosis often causes balance disturbance, cognitive decline, and reduced quality of life. Motor imagery and vestibular rehabilitation are established methods in MS care, but their effects have only been studied separately. This randomized controlled trial introduces a combined program of motor imagery and vestibular training to explore whether their integration provides broader benefits. The study will recruit patients with relapsing-remitting MS, apply an 8-week intervention, and compare outcomes in cognition, balance, physical performance, and quality of life against conventional therapy.

ELIGIBILITY:
inclusion criteria

1. Diagnosis of Multiple Sclerosis (MS) Confirmed using McDonald Criteria
2. Patient diagnosed relapsing-remitting multiple sclerosis (RRMS).
3. Mild MS between 0-3 according to PDDS.
4. Age from (18-45)
5. Mild cognitive impairment
6. Balance impairment (mild to moderate impairment)
7. Vestibular dysfunction Related to MS (dizziness, vertigo , gaze instability ) 8. Native language is Arabic to ensure clear communication during cognitive tasks and exercise instructions

9. Be able to joined the treatment (motor imagery, vestibular rehabilitaiton )

Exclusion Criteria:

Other neurological disorder, progressive multiple sclerosis Non-MS related vestibular disorders (e.g., BPPV, Meniere's disease) that would interfere with vestibular rehab.

Severe Psychiatric Conditions (schizophrenia, bipolar, etc) Sever balance disorder Sever fatigue Medical instability eg (cardiovascular disease, respiratory, infections, severe uncontrolled diabetes, or severe visual impairments.) Sever cognitive impairment Pregnant Advance disability ( wheelchair , unable to stand ) Use of Vestibular-Suppressing Medications Non - speaker Arabic

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Change in Cognitive Function (Montreal Cognitive Assessment [MoCA] Score) | Baseline and 8 weeks after intervention
  It is a cognitive screening tool commonly used in clinics and research to assess individual cognitive impairment and its severity. It helps therapists evaluate a patient's cognitive function and identify changes over time by assessing mental capacity functions and takes about 10-15 minutes to complete., which includes Attention & Concentration, Executive Functions, Memory, Language, Visuospatial Skills and Orientation (19).
  1. The test is scored out of 30 points.
  2. A score of 26 or higher is considered normal.
  3. Scores below 26 may indicate mild cognitive impairment or early dementia.
Change in Balance Berg Balance Scale [ABBS] Score) | Baseline (Week 0) and Post-intervention (Week 8)
  To assess balance and fall risk in Arabic-speaking patients with neurological disorders, lower scores indicate more severe balance problems (23).
  1. 41-56: Low fall risk, good balance.
  2. 21-40: Moderate fall risk.
  3. 0-20: High fall risk."
Change in Vestibular Function (Dynamic Visual Acuity [DVA] Test) | Baseline and Week 8.
  DVA assesses visual acuity during head movement to evaluate vestibulo-ocular reflex integrity.It is a functional test designed to evaluate the integrity of the vestibulo-ocular reflex (VOR), which stabilizes the eyes during head motion. DVA is commonly employed to detect vestibular dysfunction and is particularly useful for evaluating vestibular function in patients experiencing dizziness, balance disorders, or conditions such as multiple sclerosis (MS), where vestibular dysfunction is common
Change in Vestibular Function (Head Impulse Test [HIT]) | Baseline and Week 8
  Bedside assessment of semicircular canal/VOR function. Outcome recorded as presence/absence of corrective saccades and qualitative clinician rating of gain; improvement indicates better vestibular function.It is a clinical test used to identify deficits in the semicircular canals, especially the horizontal canal, and is useful for detecting peripheral vestibular deficits. It assesses the ability of the vestibulo-ocular reflex (VOR) to maintain stable vision during rapid, unpredictable head movements
Change in Cognitive Function (Brief International Cognitive Assessment for MS [BICAMS] Composite Score | Baseline (Week 0) and Post-intervention (Week 8)
  Cognition will be assessed using BICAMS (SDMT, CVLT-II, BVMT-R). A composite and subtest scores will be calculated; This test is valdiated in Egyption dialect. It is a specialized tool designed for patients with multiple sclerosis to assess their cognitive function. It is reliable, quick, and sensitive, making it useful for both clinical settings and research. The tool focuses on cognitive domains that are commonly affected in multiple sclerosis, such as memory, speed, and learning. It includes tests like the Symbol Digit Modalities Test (SDMT), California Verbal Learning Test-II (CVLT-II), and Brief Visuospatial Memory Test-Revised (BVMT-R)
Change in balance (Timed Up and Go [TUG] Time) | Baseline and Week 8
  Seconds to stand up, walk 3 m, turn, return, and sit. Lower times indicate better mobility; ≥12 s suggests increased fall risk.
Change in Disability Status (Patient-Determined Disease Steps [PDDS] Score) | Baseline and Week 8.
  Self-reported disability (0-8); higher scores indicate greater disability.

SECONDARY OUTCOMES:
Change in Quality of Life (Multiple Sclerosis Impact Scale-29 [MSIS-29] | Baseline and Week 8.
  The Multiple Sclerosis Impact Scale-29 (MSIS-29) is a clinical tool used by patients to assess the impact of MS on their quality of life. The questionnaire consists of 29 questions and evaluates both physical and psychological well-being, helping to determine how MS affects daily life

CONTACTS AND LOCATIONS:
Overall Officials: Merve Yılmaz Menek, Assoc. Prof, Study Director — Assoc. Prof. Merve Yılmaz Menek
Locations (1):
- Gehad Salem Mohamed Mohamed Menshawi, Istanbul, Beykoz/İstanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ozgen G, Karapolat H, Akkoc Y, Yuceyar N. Is customized vestibular rehabilitation effective in patients with multiple sclerosis? A randomized controlled trial. Eur J Phys Rehabil Med. 2016 Aug;52(4):466-78. Epub 2016 Apr 6. PMID 27050082
- [Background] Abraham A, Hart A, Andrade I, Hackney ME. Dynamic Neuro-Cognitive Imagery Improves Mental Imagery Ability, Disease Severity, and Motor and Cognitive Functions in People with Parkinson's Disease. Neural Plast. 2018 Mar 14;2018:6168507. doi: 10.1155/2018/6168507. eCollection 2018. PMID 29725348
- [Background] Aljarallah S, Alkhathlan H, Almushawah A, Badahdah A, Alfaifi N, Abdulmaged-Ahmed DA, Alkhawajah NM. Performance of an Arabic translation of the patient determined disease steps (PDDS) scale in Saudi patients with multiple sclerosis. Medicine (Baltimore). 2023 Nov 3;102(44):e35889. doi: 10.1097/MD.0000000000035889. PMID 37932990
- [Background] Rahman TT, El Gaafary MM. Montreal Cognitive Assessment Arabic version: reliability and validity prevalence of mild cognitive impairment among elderly attending geriatric clubs in Cairo. Geriatr Gerontol Int. 2009 Mar;9(1):54-61. doi: 10.1111/j.1447-0594.2008.00509.x. PMID 19260980
- [Background] Manago MM, Schenkman M, Berliner J, Hebert JR. Gaze stabilization and dynamic visual acuity in people with multiple sclerosis. J Vestib Res. 2016;26(5-6):469-477. doi: 10.3233/VES-160593. PMID 28262642
- [Background] Mulder T. Motor imagery and action observation: cognitive tools for rehabilitation. J Neural Transm (Vienna). 2007;114(10):1265-78. doi: 10.1007/s00702-007-0763-z. Epub 2007 Jun 20. PMID 17579805
- [Background] Urgesi C, Moro V, Candidi M, Aglioti SM. Mapping implied body actions in the human motor system. J Neurosci. 2006 Jul 26;26(30):7942-9. doi: 10.1523/JNEUROSCI.1289-06.2006. PMID 16870739
- [Background] Volz MS, Suarez-Contreras V, Portilla AL, Fregni F. Mental imagery-induced attention modulates pain perception and cortical excitability. BMC Neurosci. 2015 Mar 15;16:15. doi: 10.1186/s12868-015-0146-6. PMID 25887060
- [Background] Khan F, Amatya B. Rehabilitation in Multiple Sclerosis: A Systematic Review of Systematic Reviews. Arch Phys Med Rehabil. 2017 Feb;98(2):353-367. doi: 10.1016/j.apmr.2016.04.016. Epub 2016 May 20. PMID 27216225
- [Background] Efendi H. Clinically Isolated Syndromes: Clinical Characteristics, Differential Diagnosis, and Management. Noro Psikiyatr Ars. 2015 Dec;52(Suppl 1):S1-S11. doi: 10.5152/npa.2015.12608. Epub 2015 Dec 1. PMID 28360754
- [Background] McGinley MP, Goldschmidt CH, Rae-Grant AD. Diagnosis and Treatment of Multiple Sclerosis: A Review. JAMA. 2021 Feb 23;325(8):765-779. doi: 10.1001/jama.2020.26858. PMID 33620411
- [Background] Habbestad A, Willumsen JS, Aarseth JH, Grytten N, Midgard R, Wergeland S, Myhr KM, Torkildsen O. Increasing age of multiple sclerosis onset from 1920 to 2022: a population-based study. J Neurol. 2024 Apr;271(4):1610-1617. doi: 10.1007/s00415-023-12047-9. Epub 2023 Dec 14. PMID 38097800
- [Background] Walton C, King R, Rechtman L, Kaye W, Leray E, Marrie RA, Robertson N, La Rocca N, Uitdehaag B, van der Mei I, Wallin M, Helme A, Angood Napier C, Rijke N, Baneke P. Rising prevalence of multiple sclerosis worldwide: Insights from the Atlas of MS, third edition. Mult Scler. 2020 Dec;26(14):1816-1821. doi: 10.1177/1352458520970841. Epub 2020 Nov 11. PMID 33174475
- [Result] Garcia-Munoz C, Cortes-Vega MD, Heredia-Rizo AM, Martin-Valero R, Garcia-Bernal MI, Casuso-Holgado MJ. Effectiveness of Vestibular Training for Balance and Dizziness Rehabilitation in People with Multiple Sclerosis: A Systematic Review and Meta-Analysis. J Clin Med. 2020 Feb 21;9(2):590. doi: 10.3390/jcm9020590. PMID 32098162
- See also: Clinical characteristics of patients with multiple sclerosis enrolled in a new registry in Egypt — https://pubmed.ncbi.nlm.nih.gov/27919495/
- See also: Multiple Sclerosis: Pathogenesis, Symptoms, Diagnoses and Cell-Based Therapy — https://pubmed.ncbi.nlm.nih.gov/28367411/
- See also: Review of multiple sclerosis: Epidemiology, etiology, pathophysiology, and treatment — https://pubmed.ncbi.nlm.nih.gov/38394496/
- See also: Book Multiple Sclerosis Rehabilitation From Impairment to Participation Edited ByMarcia Finlayson — https://www.taylorfrancis.com/books/edit/10.1201/b12666/multiple-sclerosis-rehabilitation-marcia-finlayson
- See also: Effectiveness of Motor Imagery on Motor Recovery in Patients with Multiple Sclerosis: Systematic Review — https://pubmed.ncbi.nlm.nih.gov/33435410/
- See also: The Effectiveness of Vestibular Rehabilitation on Balance Related Impairments among Multiple Sclerosis Patients: A Systematic Review — https://www.iomcworld.org/open-access/the-effectiveness-of-vestibular-rehabilitation-on-balance-related-impairments-among-multiple-sclerosis-patients-a-systematic-revie-53345.html
- See also: Motor imagery in multiple sclerosis: exploring applications in therapeutic treatment — https://pubmed.ncbi.nlm.nih.gov/30207860/
- See also: Effectiveness of Vestibular Training for Balance and Dizziness Rehabilitation in People with Multiple Sclerosis: A Systematic Review and Meta-Analysis — https://pubmed.ncbi.nlm.nih.gov/32098162/
- See also: Vestibular Rehabilitation — https://www.ncbi.nlm.nih.gov/books/NBK572153/
- See also: Reliability and validity of Arabic version of the brief international cognitive assessment for multiple sclerosis: Egyptian dialect — https://ejnpn.springeropen.com/articles/10.1186/s41983-021-00303-6
- See also: Advances in dynamic visual acuity test research — https://www.frontiersin.org/journals/neurology/articles/10.3389/fneur.2022.1047876/full
- See also: Validation of the Arabic version of the Berg Balance Scale (A-BBS) among elderly residents in a rural community — https://www.researchgate.net/publication/275642108_Validation_of_the_Arabic_version_of_the_Berg_Balance_Scale_A-BBS_among_elderly_residents_in_a_rural_community
- See also: The reliability and validity of the Timed Up and Go as a clinical tool in individuals with and without disabilities across a lifespan: a systematic review — https://pubmed.ncbi.nlm.nih.gov/31656104/
- See also: Validation of the Arabic Version of the Multiple Sclerosis Impact Scale (MSIS-29): a Rasch Analysis Study — https://pubmed.ncbi.nlm.nih.gov/39727197/
- See also: Combined upper limb and breathing exercise programme for pain management in ambulatory and non-ambulatory multiple sclerosis individuals: part II analyses from feasibility study — https://pubmed.ncbi.nlm.nih.gov/31422507/
- See also: Exercise and multiple sclerosis — https://pubmed.ncbi.nlm.nih.gov/15575796/
- See also: Best practice for motor imagery: a systematic literature review on motor imagery training elements in five different disciplines — https://bmcmedicine.biomedcentral.com/articles/10.1186/1741-7015-9-75#citeas
- See also: Effects of Motor Imagery Training on Balance and Gait in Older Adults: A Randomized Controlled Pilot Study — https://pubmed.ncbi.nlm.nih.gov/33466699/
- See also: Rehabilitation to improve gaze and postural stability in people with multiple sclerosis: study protocol for a prospective randomized clinical trial — https://bmcneurol.biomedcentral.com/articles/10.1186/s12883-019-1353-z#citeas
- See also: Vestibular rehabilitation in multiple sclerosis: study protocol for a randomised controlled trial and cost-effectiveness analysis comparing customised with booklet based vestibular rehabilitation for vestibulopathy and a 12 month observational cohort stu — https://pubmed.ncbi.nlm.nih.gov/33243182/
- See also: Exercises for multiple sclerosis : a safe and effective program to fight fatigue, build strength, and improve balance — https://levittown-nls.na.iiivega.com/search/card?id=db4b0e0a-e0b6-5a85-8776-5fd2b5ecd6b1&entityType=FormatGroup